CLINICAL TRIAL: NCT05753449
Title: Burst-Type Deep Brain Stimulation of the Subthalamic Nucleus in Parkinson's Disease: A Pilot Study of Tolerability and Efficacy
Brief Title: Burst-Type Deep Brain Stimulation of the Subthalamic Nucleus in Parkinson's Disease
Acronym: BURST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment Challenges due to the reluctance of patients who have achieved successful outcomes with their DBS and hesitation to change their device settings.
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Nestor Tomycz, Neurosurgeon, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-234
Record Dates: First submitted 2023-02-07; First posted 2023-03-03 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind cross-over study
Who Masked: Participant, Investigator
Masking Description: Subjects will be programmed to both settings over the course of the visits, but the order is randomized to ensure appropriate blinding of the UPDRS assessor.
  Unblinded examiner will then turn the DBS ON to the patient's baseline DBS settings continuously ON or to burst DBS mode.
  A blinded examiner who did not perform the programming change will perform a UPDRS-III evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Baseline Programming First, Then Experimental Burst-type Programming (Experimental): In this arm, patients were randomized to initially receive treatment with baseline DBS programming (standard of care) at Visit 1. After a 30 minute treatment period, patients were to undergo UPDRS III evaluation, a 15 minute washout period with the DBS turned off and then experimental Burst-type programming for 30 minutes. Finally, patients were to undergo UPDRS III evaluation after the second round of programming.
  Interventions: Device: Baseline (or standard of care) DBS programming; Device: Burst-type DBS electrical stimulation programming
- Experimental Burst-type Programming First, Then Baseline Programming (Experimental): In this arm, patients were randomized to initially receive treatment with experimental Burst-type DBS programming at Visit 1. After a 30 minute treatment period, patients were to undergo UPDRS III evaluation, a 15 minute washout period with the DBS turned off and then baseline programming (standard of care) for 30 minutes. Finally, patients were to undergo UPDRS III evaluation after the second round of programming. Burst-type DBS is defined as a novel stimulation protocol in which intermittent bursts of traditional high-frequency rectangular wave stimulation are delivered.
  Interventions: Device: Baseline (or standard of care) DBS programming; Device: Burst-type DBS electrical stimulation programming

INTERVENTIONS:
Device: Baseline (or standard of care) DBS programming — Baseline (or standard of care) DBS programming.
  Other Names: Boston Scientific Neuromodulation (BSN) Vercise™ System
Device: Burst-type DBS electrical stimulation programming — Burst-type DBS is defined as a novel stimulation protocol in which intermittent bursts of traditional high-frequency rectangular wave stimulation are delivered.
  Other Names: Boston Scientific Neuromodulation (BSN) Vercise™ System

SUMMARY:
This is a study to evaluate Deep brain stimulation (DBS) burst-type electrical stimulation programming verses standard DBS programming. Burst-type DBS is defined as a novel stimulation protocol in which intermittent bursts of traditional high-frequency rectangular wave stimulation are delivered. Burst type DBS may improve the efficacy and durability of DBS pulse generator.

DETAILED DESCRIPTION:
Five (N = 5) subjects that have bilateral subthalamic nucleus deep brain stimulation (STN-DBS), with Boston Scientific Gevia or Genus technology, implanted for Parkinson's Disease (PD). Subjects should be on stable DBS programming settings and stable medication regimens defined as no DBS programming changes or Parkinson's disease medication changes over the past 2 weeks. The DBS implantation should have been performed by either Dr. Nestor D. Tomycz MD or Dr. Donald M. Whiting MD at Allegheny General Hospital and implantation surgery must have occurred a minimum of 6 months prior to the day of enrollment.

Screening Visit- All interested patients will undergo a screening visit during which their eligibility into the study will be determined. Screening will including the following:

* Review and signing of informed consent document.
* Demographics: Date of birth, Gender, Ethnicity, Handedness
* Medical history: Surgical/Interventional Procedure History, Parkinson's Disease History (presence of symptoms required for eligibility will be documented), presence and in some cases severity of selected symptoms of either PD or PD medications that can also occur as a side effect of STN-DBS dopamine dysregulation syndrome (DDS);
* Review of current Parkinson's disease medications: Dosage/frequency (Start Date, Stop Date)
* Review of concomitant medications

Visit 1- Baseline (less than or equal to 30 days after Screening

* Parkinson's disease dopaminergic medications will be withdrawn overnight to establish medication-OFF state and DBS will be turned OFF overnight for establishing DBS-OFF state. Examiner will establish a UPDRS-III baseline with medication-OFF, DBS-OFF state.
* Unblinded examiner will then turn the DBS ON to the patient's baseline DBS settings continuously ON or to burst DBS mode (baseline DBS settings for the patient with DBS set to 1 sec ON, 4 sec OFF), based on results of randomization. The patient will be blinded to this programming change and will be kept at this initial setting for 30 minutes.
* Next, a blinded examiner who did not perform the programming change will perform a UPDRS-III evaluation. Next, the DBS will be turned off for 15 minutes to permit for a washout period.
* Next, the DBS will be turned on by the unblinded examiner to the alternate setting (burst DBS in case that the patient first was turned on with their baseline DBS setting or baseline DBS setting in case that the patient was first turned on with burst DBS setting) and kept on this setting for 30 minutes.
* After 30 minutes, the blinded examiner will perform another UPDRS-III evaluation. Patients, who are blinded to the stimulation setting, will be asked if they preferred one stimulation mode over the other.
* If any adverse events occur with burst DBS mode, the unblinded examiner will decrease the amplitude of the DBS by 0.5 milliamp (mA) increments until the adverse events abate. If there are not persistent adverse events with 30 minutes of burst DBS mode, the patient will be kept in burst DBS mode at the end of first visit and will be allowed to take their Parkinson's disease medications.

Randomization- Subjects will be randomized to determine which DBS setting is initially programmed during visit one. All subjects will be programmed to both settings over the course of the visit, but the order is randomized to ensure appropriate blinding of the UPDRS assessor. Subjects have a 50% chance of being randomized to the "burst" mode, and a 50% chance of being randomized to the "baseline" mode.

Visit Two (6 months +/- 30 Days)

* Parkinson's disease dopaminergic medications will be withdrawn overnight to establish medication-OFF state and DBS will be turned OFF overnight for establishing DBS-OFF state.
* Examiner will establish a UPDRS-III baseline with medication-OFF, DBS-OFF state. Examiner will then turn the DBS ON to the burst DBS state and keep ON for 30 minutes. After 30 minutes the examiner will perform another UPDRS-III evaluation and will ask about any adverse effects. Patients will then be allowed to take their Parkinson's disease medications and will be kept on the burst mode DBS state.
* Patients will be asked if they prefer the burst mode DBS state to their baseline settings before the study.

Visit Three (12 months +/- 30 days)

* Parkinson's disease dopaminergic medications will be withdrawn overnight to establish medication-OFF state and DBS will be turned OFF overnight for establishing DBS-OFF state.
* Examiner will establish a UPDRS-III baseline with medication-OFF, DBS-OFF state. Examiner will then turn the DBS ON to the burst DBS state and keep ON for 30 minutes. After 30 minutes the examiner will perform another UPDRS-III evaluation and will ask about any adverse effects. Patients will then be allowed to take their Parkinson's disease medications and will be kept on the burst mode DBS state.
* Patients will be asked if they prefer the burst mode DBS state to their baseline settings before the study. At the conclusion of the study, patients will be asked if they want to continue to use burst DBS state or if would prefer to be programmed back to their pre-study baseline DBS settings.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral DBS-STN (subthalamic nucleus) target for idiopathic Parkinson's disease implanted minimum 6 months prior to the day of study enrollment
* Stable DBS programming settings and Parkinson's disease medications defined as no changes to either within past 2 weeks
* Comfortable using DBS controller to turn off device prior to study visits
* Able to provide informed consent and complete follow-up visits

Exclusion Criteria:

* DBS technology other than Boston scientific Genus/Gevia
* Unable to complete follow-up visits
* DBS brain targets other than STN (subthalamic nucleus)
* Signs of progressive cognitive decline

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Tomycz, Principal Investigator — Allegheny Health Network AGH Department of Neuroscience
Locations (1):
- AHN Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 subjects were recruited in the medical clinic between August 24, 2022, and February 21, 2024. Recruitment ended as we encountered significant challenges in recruiting participants for the study finding reluctance of patients who have achieved successful outcomes with their deep brain stimulation (DBS) devices to participate. They are understandably hesitant to risk potential symptom worsening by altering their device settings, even for the purpose of research.
Period: Visit 1: First Treatment (30 Min)
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming
Started | 0 (No subjects were randomized to this arm.) | 2
Completed | 0 (No subjects were randomized to this arm.) | 2
Not Completed | 0 | 0
Period: Visit 1: Washout Period (15 Min)
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming
Started | 0 (No subjects were randomized to this arm.) | 2
Completed | 0 (No subjects were randomized to this arm.) | 2
Not Completed | 0 | 0
Period: Visit 1: Second Treatment (30 Min)
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming
Started | 0 (No subjects were randomized to this arm.) | 2
Completed | 0 (No subjects were randomized to this arm.) | 2
Not Completed | 0 | 0
Period: Visit 2: Burst-type Programming (30 Min)
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming
Started | 0 (No subjects were randomized to this arm.) | 1 (One subject in this arm dropped out from the study prior to Visit 2.)
Completed | 0 (No subjects were randomized to this arm.) | 1 (One subject in this arm dropped out from the study prior to Visit 2.)
Not Completed | 0 | 0
Period: Visit 3: Burst-type Programming (30 Min)
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming
Started | 0 (No subjects were randomized to this arm.) | 1 (One subject in this arm dropped out from the study prior to Visit 2.)
Completed | 0 (No subjects were randomized to this arm.) | 1 (One subject in this arm dropped out from the study prior to Visit 2.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were enrolled in the standard of care programming arm. 2 were enrolled in the Experimental/Burst type programming arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] |  | 70 [65 to 75] | 70 [65 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) v-III Motor Examination Scores at Baseline (Visit 1)
Description: This outcome is the Unified Parkinson's Disease Rating Scale (UPDRS) v-III Motor Examination Score in the "Medication Off" state, after the first treatment (administered for 30 minutes) and after the second treatment (administered for 30 minutes). For example, the first treatment for patients in the arm "Baseline Programming First, Then Experimental Burst-type Programming" was baseline (or standard of care) DBS programming, and the second treatment was experimental Burst-style programming. Each item is scored on a scale from 0 (normal) to 4 (severe, marked, or unable), with the total possible score for the 14 items, including separate questions regarding symptoms present axially and in appendages, ranging from 0 to 108. A higher score indicates a worse outcome.
Time Frame: Baseline
Population: No subjects were randomized to the arm that received baseline (standard of care) programming first, followed by experimental Burst-style programming (at Visit 1).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming | Experimental Burst-type Programming First, Then Baseline Programming
Number analyzed (Participants) | 0 | 2
score on a scale
  Medication-Off and DBS-Off State |  | 55.5 [33 to 78]
  First Treatment / Programming Setting |  | 20 [18 to 22]
  Second Treatment / Programming Setting |  | 32 [22 to 42]

2. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) v-III Motor Examination Scores at Six Months (Visit 2)
Description: This outcomes is the Unified Parkinson's Disease Rating Scale (UPDRS) v-III Motor Examination Score in the "Medication Off" state and after burst-type DBS programming in the acute setting (after 30 minutes) at six months. Each item is scored on a scale from 0 (normal) to 4 (severe, marked, or unable), with the total possible score for the 14 items, including separate questions regarding symptoms present axially and in appendages, ranging from 0 to 108. A higher score means a worse outcome. Note that the study arm titles refer to whether or not the patients were randomized to baseline programming or Burst-type programming at Visit 1. During this visit (Visit 2), all study subjects were to be evaluated in the medication-off state and then evaluated following 30 minutes of treatment with Burst-type programming. Treatment with baseline programming was not administered during this visit (Visit 2).
Time Frame: 6 months
Population: No subjects were randomized to the arm that received baseline (standard of care) programming first, followed by experimental Burst-style programming (at Visit 1). Follow-up data at six months (Visit 2) were only available for one of the two patients randomized to first be treated with the experimental Burst-type programming at Visit 1. Additionally, data were not collected in the Medication Off state for the patient for whom there are follow-up data at six months (Visit 2).
Measure: Median (Full Range); unit: score on a scale
Groups:
- Baseline Programming First, Then Experimental Burst-type Programming (at Visit 1): In this arm, patients were randomized to initially receive treatment with baseline DBS programming (standard of care) at Visit 1. After a 30 minute treatment period, patients were to undergo UPDRS III evaluation, a 15 minute washout period with the DBS turned off and then experimental Burst-type programming for 30 minutes. Finally, patients were to undergo UPDRS III evaluation after the second round of programming.
- Experimental Burst-type Programming First, Then Baseline Programming (at Visit 1): In this arm, patients were randomized to initially receive treatment with experimental Burst-type DBS programming at Visit 1. After a 30 minute treatment period, patients were to undergo UPDRS III evaluation, a 15 minute washout period with the DBS turned off and then baseline programming (standard of care) for 30 minutes. Finally, patients were to undergo UPDRS III evaluation after the second round of programming. Burst-type DBS is defined as a novel stimulation protocol in which intermittent bursts of traditional high-frequency rectangular wave stimulation are delivered.
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming (at Visit 1) | Experimental Burst-type Programming First, Then Baseline Programming (at Visit 1)
Number analyzed (Participants) | 0 | 1
score on a scale
  Medication-Off and DBS-Off State: number analyzed (Participants) | 0 | 0
  Burst-type Programming |  | 25 [25 to 25]

3. Primary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) v-III Motor Examination Scores at Twelve Months (Visit 3)
Description: This outcomes is the Unified Parkinson's Disease Rating Scale (UPDRS) v-III Motor Examination Score in the "Medication Off" state and after burst-type DBS programming in the acute setting (after 30 minutes) at 12 months. Each item is scored on a scale from 0 (normal) to 4 (severe, marked, or unable), with the total possible score for the 14 items, including separate questions regarding symptoms present axially and in appendages, ranging from 0 to 108. A higher score means a worse outcome. Note that the study arm titles refer to whether or not the patients were randomized to baseline programming or Burst-type programming at Visit 1. During this visit (Visit 2), all study subjects were to be evaluated in the medication-off state and then evaluated following 30 minutes of treatment with Burst-type programming. Treatment with baseline programming was not administered during this visit (Visit 2).
Time Frame: 12 months
Population: No subjects were randomized to the arm that received baseline (standard of care) programming first, followed by experimental Burst-style programming (at Visit 1). Follow-up data at 12 months were only available for one of the two patients randomized to first be treated with the experimental Burst-type programming at Visit 1. Additionally, data were not collected in the Medication Off state for the patient for whom there are follow-up data at six months (Visit 2).
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming (at Visit 1) | Experimental Burst-type Programming First, Then Baseline Programming (at Visit 1)
Number analyzed (Participants) | 0 | 1
score on a scale
  Medication-Off and DBS-Off State: number analyzed (Participants) | 0 | 0
  Burst-type Programming |  | 26 [26 to 26]

ADVERSE EVENTS:
Time Frame: 364 Days
Description: While this study has been entered as a cross-over study, the only cross-over element of the study occurred during Visit 1. Because of this, the short duration of the treatment periods (of 30 minutes) and the washout period (of 15 minutes) during this visit and the possibility of adverse events in between study visits, adverse events were summarized for the entire study duration and not by treatment period on Visit 1. No adverse events occurred.
Arm/Group | Baseline Programming First, Then Experimental Burst-type Programming (at Visit 1) | Experimental Burst-type Programming First, Then Baseline Programming (at Visit 1)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
This study was terminated due to challenges in recruiting participants as reluctance of patients who have achieved successful outcomes with their DBS devices to participate. They are understandably hesitant to risk potential symptom worsening by altering their device settings, even for the purpose of research. One subject completed the trial and the second subject withdrew due to intolerance of the device settings. Both subjects were enrolled in the experimental arm of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/49/NCT05753449/Prot_SAP_000.pdf